CLINICAL TRIAL: NCT01505166
Title: Randomized Phase II Trial of Post-operative Adjuvant Chemotherapy ± FANG™ Autologous Tumor Cell Vaccine in Colorectal Carcinoma With Liver Metastases
Brief Title: Randomized Phase II Adjuvant Chemotherapy ± FANG™ in Colorectal Carcinoma With Liver Metastases
Acronym: FANG-CLM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated (Business Decision to pursue other indications)
Sponsor: Gradalis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CL-PTL 107
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Colon Cancer
Keywords: colorectal carcinoma; colon cancer; liver metastases
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vigil™ (Experimental): Patients will receive 1 x 10^7 cells (Group A) via intradermal injection for a minimum of 4 doses and a maximum of 12 doses (vaccine) starting post-surgery Week 4-8 (C1W1D1) and continuing C1W3D1, C2W3D1, then every 28 days.
  Interventions: Biological: Vigil™ Vaccine
- Placebo (Placebo Comparator): Patients will receive placebo (Group B) via intradermal injection for a minimum of 4 doses and a maximum of 12 doses starting post-surgery Week 4-8 (C1W1D1) and continuing C1W3D1, C2W3D1, then every 28 days.
  Interventions: Drug: Placebo
- Vigil™ Vaccine (6 patient run-in) (Experimental): Six patients will be enrolled into the Part 1 of the study to receive intradermal autologous Vigil™ cancer vaccine (1.0 x 10e7 cells/injection; maximum of 12 vaccinations).
  Interventions: Biological: Vigil™ Vaccine

INTERVENTIONS:
Biological: Vigil™ Vaccine — Patients will receive 1 x 10^7 cells (Group A) or placebo (Group B) via intradermal injection for a minimum of 5 doses and a maximum of 12 doses starting post-surgery Week 4-8 (C1W1D1) and continuing C1W3D1, C2W3D1, then every 28 days. Starting C1W4D1, all patients will receive modified FOLFOX6 (oxaliplatin 85 mg/m2 D1, l-leucovorin 200 mg/m2 D1, fluorouracil 400 mg/m2 IV bolus (or short infusion) D1, fluorouracil 2400 mg/m2 46 hours continuous infusion every 14 days x 6 cycles (1 cycle = 4 weeks).
  Other Names: formerly known as FANG™
  Arms: Vigil™; Vigil™ Vaccine (6 patient run-in)
Drug: Placebo — Patients will receive 1 x 10^7 cells (Group A) or placebo (Group B) via intradermal injection for a minimum of 5 doses and a maximum of 12 doses starting post-surgery Week 4-8 (C1W1D1) and continuing C1W3D1, C2W3D1, then every 28 days. Starting C1W4D1, all patients will receive modified FOLFOX6 (oxaliplatin 85 mg/m2 D1, l-leucovorin 200 mg/m2 D1, fluorouracil 400 mg/m2 IV bolus (or short infusion) D1, fluorouracil 2400 mg/m2 46 hours continuous infusion every 14 days x 6 cycles (1 cycle = 4 weeks).
  Arms: Placebo

SUMMARY:
Preliminary studies with a variety of vaccines suggest target accessibility (potential immunogenicity) in a variety of solid tumors to immune directed approaches. In an effort to overcome limitations of immunostimulatory cancer vaccines, Gradalis has designed a novel autologous vaccine to address inability to fully identify cancer associated antigens, antigen recognition by the immune system (i.e. antigen-->immunogen), effector potency, and cancer-induced resistance. In an effort to overcome limitations of immunostimulatory cancer vaccines, we designed a novel dual-modulatory autologous whole cell vaccine, Vigil™, incorporating the rhGMCSF transgene and the bifunctional shRNAfurin (to block proprotein conversion to active TGFb1 and b2) to 1) address the inability to fully identify cancer associated antigens, 2) effect antigen recognition by the immune system, 3) enhance effector potency, and 4) subvert endogenous cancer-induced immune resistance. We have also completed the Phase I assessment of Vigil™ vaccine in 30 advanced solid tumor patients (1.0 x 10^7 cells/injection/month for a maximum of 12 vaccinations) who have not experienced any significant adverse effects following 144 vaccinations, including 6 patients with colorectal carcinoma. Plasmid functionality, immune biomarker response, and preliminary evidence of anticancer activity have been observed. This is a two-part Phase II study of the Vigil™ autologous vaccine. Six patients will be enrolled into the Part 1 of the study to receive intradermal autologous Vigil™ cancer vaccine (1.0 x 10^7 cells/injection; maximum of 12 vaccinations). Part 2 of the study will be a randomized Phase II study of sandwich or adjuvant chemotherapy and intradermal autologous Vigil™ cancer vaccine (1.0 x 10^7 cells/injection; maximum of 12 vaccinations) versus sandwich or adjuvant chemotherapy and placebo in patients with colorectal carcinoma with either synchronous or metachronous liver metastases (CLM +/= pulmonary metastases) following resection +/= ablation with curative intent.Sandwich therapy indicates a combination of both pre-operative and postoperative chemotherapy as opposed to neo-adjuvant (all chemotherapy prior to surgery) or adjuvant (all chemotherapy following surgery) therapy. A minimum harvest aliquot to produce 4 monthly injections will be required for entry into the study. Patients in whom insufficient tissue (<4 doses) is collected or whose vaccine fails manufacturing release criteria will not receive vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colorectal carcinoma with synchronous or metachronous liver metastases +/- pulmonary metastases.
2. Part 1 patients: May have multiple number of metastatic lesions as long as they can be rendered no evidence of disease (NED).
3. Part 2 patients: Maximum total number of metastatic lesions </= 6. (Patients with CLM with EHD other than lung will be evaluated on an individual basis by the sponsor).

   1. For patients with 1 but up to 3 total lesions, distribution must include both liver + pulmonary metastases.
   2. For patients with 4-6 total lesions, distribution may include liver +/- pulmonary metastases.
4. Candidate for surgical excision +/= ablation with curative intent based on pre-operative assessment incorporating a CT/PET scan.
5. Has been informed of all alternative ≥ first and/or second-line therapies that are the current standard of care. If no conventional frontline therapy indicated or acceptable by patient, patient may participate after review by sponsor.
6. Planned resected viable tumor in sufficient quantity ("golf ball size" estimated weight ~ 30 grams) for vaccine processing.
7. Recovered to ≤ Grade 1 (excluding alopecia) from all clinically relevant toxicities related to prior therapies.
8. Patients must be off all "statin" drugs for ≥ 2 weeks prior to initiation of therapy.
9. Age ≥18 years.
10. ECOG performance status (PS) 0-2.
11. Estimated >4 month survival probability.
12. Normal organ and marrow function as defined below:

    Absolute granulocyte count ≥1,500/mm3 Absolute lymphocyte count ≥ 500/mm3 Platelets ≥100,000/mm3 Total bilirubin </=2 mg/dL AST(SGOT)/ALT(SGPT) </=2x institutional upper limit of normal Creatinine <1.5 mg/dL
13. Ability to understand and the willingness to sign a written informed consent document.
14. Negative pregnancy test.

Exclusion Criteria:

1. Surgery involving general anesthesia, radiotherapy, steroid therapy, or immunotherapy within 4 weeks prior to entering the study. Collection of lumenal tissue must be avoided.
2. Prior therapeutic chemotherapy (excluding protocol defined sandwich chemotherapy). Prior approved sandwich / adjuvant therapy is permitted maximum of 3 cycles (1 cycle = 2 biweekly courses / 1 month) anterior therapy and at least 6 months between cessation of chemotherapy and the diagnosis of metastatic disease.
3. Prior surgical resection, ablation or radiation therapy for metastatic disease prior to or at the time of tissue procurement.
4. Portal, celiac or periaortic metastases.
5. Patient must not have received any other investigational agents within 30 days prior to study entry/ registration.
6. Patients with known active or symptomatic brain metastases.
7. Patients with compromised pulmonary disease.
8. Short term (<30 days) concurrent systemic steroids ≤ 0.125 mg/kg prednisone per day (maximum 10 mg/day) and bronchodilators (inhaled steroids) are permitted; other steroid regimens and/or immunosuppressives are excluded.
9. Prior splenectomy.
10. Prior malignancy (excluding nonmelanoma carcinomas of the skin) unless in remission for ≥ 2 years.
11. Kaposi's Sarcoma.
12. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
13. Patients with known HIV.
14. Patients with chronic Hepatitis B and C infection.
15. Patients with uncontrolled autoimmune diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minal Barve, MD, Principal Investigator — Mary Crowley Cancer Research Centers
Locations (1):
- Mary Crowley Cancer Research Centers, Dallas, Texas, United States

REFERENCES:
- [Background] Ghisoli M, Barve M, Schneider R, Mennel R, Lenarsky C, Wallraven G, Pappen BO, LaNoue J, Kumar P, Nemunaitis D, Roth A, Nemunaitis J, Whiting S, Senzer N, Fletcher FA, Nemunaitis J. Pilot Trial of FANG Immunotherapy in Ewing's Sarcoma. Mol Ther. 2015 Jun;23(6):1103-1109. doi: 10.1038/mt.2015.43. Epub 2015 Mar 19. PMID 25917459
- [Background] Senzer N, Barve M, Kuhn J, Melnyk A, Beitsch P, Lazar M, Lifshitz S, Magee M, Oh J, Mill SW, Bedell C, Higgs C, Kumar P, Yu Y, Norvell F, Phalon C, Taquet N, Rao DD, Wang Z, Jay CM, Pappen BO, Wallraven G, Brunicardi FC, Shanahan DM, Maples PB, Nemunaitis J. Phase I trial of "bi-shRNAi(furin)/GMCSF DNA/autologous tumor cell" vaccine (FANG) in advanced cancer. Mol Ther. 2012 Mar;20(3):679-86. doi: 10.1038/mt.2011.269. Epub 2011 Dec 20. PMID 22186789
- [Background] Nemunaitis J, Barve M, Orr D, Kuhn J, Magee M, Lamont J, Bedell C, Wallraven G, Pappen BO, Roth A, Horvath S, Nemunaitis D, Kumar P, Maples PB, Senzer N. Summary of bi-shRNA/GM-CSF augmented autologous tumor cell immunotherapy (FANG) in advanced cancer of the liver. Oncology. 2014;87(1):21-9. doi: 10.1159/000360993. Epub 2014 Jun 25. PMID 24968881
- [Background] Ghisoli M, Barve M, Mennel R, Lenarsky C, Horvath S, Wallraven G, Pappen BO, Whiting S, Rao D, Senzer N, Nemunaitis J. Three-year Follow up of GMCSF/bi-shRNA(furin) DNA-transfected Autologous Tumor Immunotherapy (Vigil) in Metastatic Advanced Ewing's Sarcoma. Mol Ther. 2016 Aug;24(8):1478-83. doi: 10.1038/mt.2016.86. Epub 2016 Apr 25. PMID 27109631
- [Background] Ghisoli M, Rutledge M, Stephens PJ, Mennel R, Barve M, Manley M, Oliai BR, Murphy KM, Manning L, Gutierrez B, Rangadass P, Walker A, Wang Z, Rao D, Adams N, Wallraven G, Senzer N, Nemunaitis J. Case Report: Immune-mediated Complete Response in a Patient With Recurrent Advanced Ewing Sarcoma (EWS) After Vigil Immunotherapy. J Pediatr Hematol Oncol. 2017 May;39(4):e183-e186. doi: 10.1097/MPH.0000000000000822. PMID 28338569
- [Background] Oh J, Barve M, Matthews CM, Koon EC, Heffernan TP, Fine B, Grosen E, Bergman MK, Fleming EL, DeMars LR, West L, Spitz DL, Goodman H, Hancock KC, Wallraven G, Kumar P, Bognar E, Manning L, Pappen BO, Adams N, Senzer N, Nemunaitis J. Phase II study of Vigil(R) DNA engineered immunotherapy as maintenance in advanced stage ovarian cancer. Gynecol Oncol. 2016 Dec;143(3):504-510. doi: 10.1016/j.ygyno.2016.09.018. Epub 2016 Sep 24. PMID 27678295
- [Result] Long-term followup of bi-shRNAfurin and GMCSF augmented autologous tumor cell immunotherapy treated colorectal cancer patients in phase I and IIa studies. Minal A. Barve, Anton M. Melnyk, Luisa Manning, Gladice Wallraven, Martin Birkhofer, and John J. Nemunaitis Journal of Clinical Oncology 2017 35:15_suppl, e15100-e15100
- [Result] Barve V, Adams N, Stanbery L, Manning L, Horvath S, Wallraven G, Bognar E, Barve M, Nemunaitis J. Case Report: Marked Survival Advantage of Two Colorectal Cancer Patients with Liver Metastases Treated with Vigil and FOLFOX-6. Vaccines (Basel). 2021 Oct 18;9(10):1201. doi: 10.3390/vaccines9101201. PMID 34696309

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited patients with colorectal carcinoma with liver metastases following resection and had successful manufacturing of Vigil (minimum of 4 doses). Part 1 would enroll the first 6 patients (Vigil plus chemotherapy) and then Part 2 would randomize subsequent patients (Vigil plus chemotherapy or Placebo plus chemotherapy).
Pre-assignment Details: 3 subjects were enrolled in Part 1 and completed Vigil plus chemotherapy. No other subjects were enrolled in Part 1 and also Part 2.
Groups:
- Vigil™ Vaccine (Part 1) - 6 Patient run-in: Six patients will be enrolled into the Part 1 of the study to receive intradermal autologous Vigil™ cancer vaccine (1.0 x 10e7 cells/injection; maximum of 12 vaccinations).
  Vigil™ Vaccine: Patients will receive 1 x 10^7 cells (Group A) or placebo (Group B) via intradermal injection for a minimum of 5 doses and a maximum of 12 doses starting post-surgery Week 4-8 (C1W1D1) and continuing C1W3D1, C2W3D1, then every 28 days. Starting C1W4D1, all patients will receive modified FOLFOX6 (oxaliplatin 85 mg/m2 D1, l-leucovorin 200 mg/m2 D1, fluorouracil 400 mg/m2 IV bolus (or short infusion) D1, fluorouracil 2400 mg/m2 46 hours continuous infusion every 14 days x 6 cycles (1 cycle = 4 weeks).
- Vigil™ (Part 2): Patients will receive 1 x 10^7 cells (Group A) via intradermal injection for a minimum of 4 doses and a maximum of 12 doses (vaccine) starting post-surgery Week 4-8 (C1W1D1) and continuing C1W3D1, C2W3D1, then every 28 days.
  Vigil™ Vaccine: Patients will receive 1 x 10^7 cells (Group A) or placebo (Group B) via intradermal injection for a minimum of 5 doses and a maximum of 12 doses starting post-surgery Week 4-8 (C1W1D1) and continuing C1W3D1, C2W3D1, then every 28 days. Starting C1W4D1, all patients will receive modified FOLFOX6 (oxaliplatin 85 mg/m2 D1, l-leucovorin 200 mg/m2 D1, fluorouracil 400 mg/m2 IV bolus (or short infusion) D1, fluorouracil 2400 mg/m2 46 hours continuous infusion every 14 days x 6 cycles (1 cycle = 4 weeks).
- Placebo (Part 2): Patients will receive placebo (Group B) via intradermal injection for a minimum of 4 doses and a maximum of 12 doses starting post-surgery Week 4-8 (C1W1D1) and continuing C1W3D1, C2W3D1, then every 28 days.
  Placebo: Patients will receive 1 x 10^7 cells (Group A) or placebo (Group B) via intradermal injection for a minimum of 5 doses and a maximum of 12 doses starting post-surgery Week 4-8 (C1W1D1) and continuing C1W3D1, C2W3D1, then every 28 days. Starting C1W4D1, all patients will receive modified FOLFOX6 (oxaliplatin 85 mg/m2 D1, l-leucovorin 200 mg/m2 D1, fluorouracil 400 mg/m2 IV bolus (or short infusion) D1, fluorouracil 2400 mg/m2 46 hours continuous infusion every 14 days x 6 cycles (1 cycle = 4 weeks).
Period: Overall Study
Arm/Group | Vigil™ Vaccine (Part 1) - 6 Patient run-in | Vigil™ (Part 2) | Placebo (Part 2)
Started | 3 | 0 | 0
Completed | 3 ("Completed" means subject had successful Vigil manufacturing and had been given all the doses.) | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study closed to enrollment and Part 2 was not initiated.
Groups:
- Vigil™ Vaccine (Part 1) 6 Patient run-in: Six patients will be enrolled into the Part 1 of the study to receive intradermal autologous Vigil™ cancer vaccine (1.0 x 10e7 cells/injection; maximum of 12 vaccinations).
  Vigil™ Vaccine: Patients will receive 1 x 10^7 cells (Group A) or placebo (Group B) via intradermal injection for a minimum of 5 doses and a maximum of 12 doses starting post-surgery Week 4-8 (C1W1D1) and continuing C1W3D1, C2W3D1, then every 28 days. Starting C1W4D1, all patients will receive modified FOLFOX6 (oxaliplatin 85 mg/m2 D1, l-leucovorin 200 mg/m2 D1, fluorouracil 400 mg/m2 IV bolus (or short infusion) D1, fluorouracil 2400 mg/m2 46 hours continuous infusion every 14 days x 6 cycles (1 cycle = 4 weeks).
- Total: Total of all reporting groups
Arm/Group | Vigil™ Vaccine (Part 1) 6 Patient run-in | Vigil™ (Part 2) | Placebo (Part 2) | Total
Number analyzed (Participants) | 3 | 0 | 0 | 3
Age, Customized [Count of Participants; unit: Participants]
  0-15 Years | 0 |  |  | 0
  16-64 Years | 2 |  |  | 2
  65 Years and Older | 1 |  |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  |  | 2
  Male | 1 |  |  | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 3 |  |  | 3
  Black/African American | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Hispanic | 0 |  |  | 0
  Other | 0 |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Immune Analysis in Tumor Biopsy and Blood (Part 1)
Description: To evaluate and correlate Tumor Infiltrating Lymphocytes (TIL) in initial excised tumor and Enzyme-Linked ImmunoSorbent Spot (ELISPOT) responses to Vigil™ vaccine in blood of patients with CLM.
Time Frame: Up to 12 months
Population: 3 subjects were enrolled in Part 1 and completed Vigil plus chemotherapy. However, TIL was not tested/collected so no correlation could be performed. Statistical analysis was not done. This study was terminated.
Arm/Group | Vigil™ Vaccine (Part 1) - 6 Patient run-in
Number analyzed (Participants) | 0

2. Primary Outcome: Percent of Patients Who Progressed After Treatment (Part 2)
Description: Response rate will also be evaluated in this study using the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST) (unidimensional measurement) of the tumor lesions are used in the RECIST criteria.The response in patients with measurable disease will be reported using standard outcome measures for clinical trials: complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD). Any response to treatment (either PR or CR) requires two confirmatory staging at least 4 weeks apart. Patients will be evaluable for tumor response if measurable disease is present.
Time Frame: 24 months
Population: This outcome measure was for Part 2. No subjects were randomized in Part 2. This study was terminated.
Arm/Group | Vigil™ (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Percent of Patients Who Survived After Treatment (Part 2)
Description: To determine and compare the overall survival rate in patients with CLM following resection +/- ablation with curative intent treated with sandwich or adjuvant chemotherapy and Vigil™ vaccine versus sandwich or adjuvant chemotherapy and placebo and compare with historical data.
Time Frame: 24 months
Population: This outcome measure was for Part 2. No subjects were randomized in Part 2. This study was terminated.
Arm/Group | Vigil™ (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Enzyme-Linked ImmunoSorbent Spot (ELISPOT) (Part 1)
Description: To determine if subjects will have a positive (defined as >10 ELISPOTS from baseline) immune response to Vigil. Blood was collected to compare ELISPOT results from baseline until 30 days after last dose.
Time Frame: Baseline, End of Treatment (30 days after last dose) up to 12 months
Population: 3 subjects were enrolled in Part 1 and completed Vigil plus chemotherapy. After 12 months, all 3 subjects had positive ELISPOT response. Statistical analysis was not done. This study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | Vigil™ Vaccine (6 Patient run-in)
Number analyzed (Participants) | 3
Participants
  ELISPOT-Positive After 12 months | 3
  ELISPOT-Negative After 12 months | 0

5. Other Pre Specified Outcome: Number of Alive Subjects (Part 1)
Description: For Part 1, this was to determine the overall survival rate in patients with CLM following resection +/= ablation with curative intent treated with adjuvant chemotherapy and Vigil™ by following these patients up to 24 months.
Time Frame: 24 Months
Population: 3 subjects were enrolled in Part 1 and completed Vigil plus chemotherapy. After 24 months, 2 subjects were still alive and 1 subject was dead. Statistical analysis was not done. This study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | Vigil™ Vaccine (Part 1) 6 Patient run-in
Number analyzed (Participants) | 3
Participants
  Alive after 24 months | 2
  Dead after 24 months | 1

ADVERSE EVENTS:
Description: At the time that the trial closed, only one subject had died. The other two were still alive. Three serious adverse events were reported during the same hospitalization for one subject.
Arm/Group | Vigil™ | Placebo | Vigil™ Vaccine (6 Patient run-in)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 1/3
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vigil™ (N=0) | Placebo (N=0) | Vigil™ Vaccine (6 Patient run-in) (N=3)
Thromboembolic Event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vigil™ (N=0) | Placebo (N=0) | Vigil™ Vaccine (6 Patient run-in) (N=3)
Injection Site Reaction (General disorders) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes